CLINICAL TRIAL: NCT03869866
Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Potential Pilgrims Aged 56 Years and Older
Brief Title: Study to Assess the Safety and Immunogenicity of a Single Dose of a Quadrivalent Meningococcal Conjugate Vaccine (MenACYW Conjugate Vaccine) in Older Adults in Turkey and Lebanon
Acronym: MEQ00063
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MEQ00063; U1111-1183-6163 (Registry Identifier: ICTRP)
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers (Meningococcal Infection)
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MenACYW conjugate vaccine (Experimental): MenACYW conjugate single injection at Day 0
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid conjugate vaccine MenACYW conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid conjugate vaccine MenACYW conjugate vaccine — Pharmaceutical form: Solution for injection Route of administration: Intramuscular
  Other Names: MenQuadfi®

SUMMARY:
The primary objectives of this study are:

* To describe the antibody response to meningococcal serogroups A, C, W, and Y measured by serum bactericidal assay using baby rabbit complement (rSBA) before and after a single dose of MenACYW conjugate vaccine
* To describe the antibody response to meningococcal serogroups A, C, W, and Y measured by serum bactericidal assay using human complement (hSBA) before and after a single dose of MenACYW conjugate vaccine
* To describe the antibody responses against tetanus toxoid at baseline and after a single dose of MenACYW conjugate vaccine
* To describe the safety profile of a single dose of MenACYW conjugate vaccine

DETAILED DESCRIPTION:
Study duration per participant is approximately 30 days including: 1 day of screening and vaccination, a phone call and a safety follow up/end of study visit at Day 8 and Day 30 after vaccine administration, respectively.

ELIGIBILITY:
Inclusion criteria :

* Aged ≥ 56 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* Intending to go on a Hajj or Umrah pilgrimage (but not within the next 10 to 12 months after vaccination)

Exclusion criteria:

* Participant is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year or surgically sterile).
* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine prior to Visit 2 except for influenza vaccination, which may be received at least 2 weeks before or after study vaccine. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Any previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, B, C, W, or Y).
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia).
* Known systemic hypersensitivity to any of the vaccine components, or history of a lifethreatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances .
* Personal history of Guillain-Barre syndrome (GBS).
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine within at least 10 years of the proposed study vaccination.
* Verbal report thrombocytopenia, contraindicating intramuscular vaccination, in the Investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness (eg, human immunodeficiency virus [HIV], hepatitis B, hepatitis C) that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0 C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (3):
- Investigational Site Number : 4220001, Beirut, Lebanon
- Turkey (Türkiye) (2):
  - Investigational Site Number : 7920002, Ankara
  - Investigational Site Number : 7920001, Ankara

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Dbaibo GS, Balik I, Akdemir I, Buzgan T, Guner R, Boutros CF, Damaj S, Zein ZE, Merhi S, Faour K, Tfaily N, Khafaja S, Dogu A, Ceyhan M. Immunogenicity and Safety of Quadrivalent Meningococcal Conjugate Vaccine (MenACYW-TT) in Potential Hajj/Umrah Pilgrims Aged >/= 56 Years: A Phase III, Open-Label Study. Infect Dis Ther. 2026 Jan 28. doi: 10.1007/s40121-025-01298-w. Online ahead of print. PMID 41604139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 centers in 2 countries between 08 April 2019 to 18 March 2022.
Pre-assignment Details: A total of 290 participants who met all the inclusion criteria were enrolled in the study.
Groups:
- MenACYW Conjugate Vaccine: Participants received a single dose of meningococcal polysaccharide [Serogroups A, C, W and Y (MenACYW conjugate vaccine)] 0.5 milliliter (mL) intramuscular (IM) injection on Day 0.
Period: Overall Study
Arm/Group | MenACYW Conjugate Vaccine
Started | 290
Vaccinated (Participants who had received at least 1 dose of the study vaccine.) | 288
Completed | 286
Not Completed | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Participants with data in case report form (CRF) consisted of all study participants with CRF, i.e with data in the clinical database.
Groups:
- MenACYW Conjugate Vaccine: Participants received a single dose of meningococcal polysaccharide [Serogroups A, C, W and Y (MenACYW conjugate vaccine)] 0.5 mL IM injection on Day 0.
Arm/Group | MenACYW Conjugate Vaccine
Number analyzed (Participants) | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 188
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 290
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Baby Rabbit Complement (rSBA) Antibody Titers Greater Than or Equal to (>=) 1:8 Against Meningococcal Serogroups A, C, W, and Y
Description: Functional meningococcal antibody activity against serogroups A, C, W, and Y were measured in a serum bactericidal assay utilizing the rSBA. Seroprotection rate is defined as percentage of participants with rSBA titer >=1.8 who received MenACYW conjugate vaccine. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post-dose
Population: The Full analysis set (FAS) consisted of participants who received at least 1 dose of the study vaccine and had a valid post-vaccination serology result. Only those participants with data collected are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW Conjugate Vaccine
Number analyzed (Participants) | 287
percentage of participants
  Serogroup A: number analyzed (Participants) | 273
  Serogroup A | 90.1 [85.9 to 93.4]
  Serogroup C | 94.1 [90.7 to 96.5]
  Serogroup W | 91.3 [87.4 to 94.3]
  Serogroup Y | 95.5 [92.4 to 97.6]

2. Primary Outcome: Geometric Mean Titers Against Meningococcal Serogroups A, C, W, and Y Measured by rSBA
Description: Functional meningococcal antibody activity against serogroups A, C, W, and Y were measured in a serum bactericidal assay utilizing the rSBA and the results were expressed as geometric mean titers.
Time Frame: Day 30 post-dose
Population: The FAS consisted of participants who received at least 1 dose of the study vaccine and had a valid post-vaccination serology result. Only those participants with data collected are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenACYW Conjugate Vaccine
Number analyzed (Participants) | 287
Titer
  Serogroup A: number analyzed (Participants) | 273
  Serogroup A | 635 [477 to 845]
  Serogroup C | 2038 [1529 to 2718]
  Serogroup W | 2710 [1929 to 3807]
  Serogroup Y | 2539 [1970 to 3272]

3. Primary Outcome: Geometric Mean Titers Against Meningococcal Serogroups A, C, W, and Y Measured by Serum Bactericidal Assay Using Human Complement (hSBA)
Description: Functional meningococcal antibody activity against serogroups A, C, W, and Y were measured in a serum bactericidal assay utilizing the hSBA and the results were expressed as geometric mean titers.
Time Frame: Day 30 post-dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenACYW Conjugate Vaccine
Number analyzed (Participants) | 287
Titer
  Serogroup A | 31.9 [26.3 to 38.8]
  Serogroup C | 135 [105 to 172]
  Serogroup W | 56.3 [44.0 to 72.1]
  Serogroup Y | 130 [102 to 165]

4. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies Against Tetanus Toxoid
Description: Tetanus toxoid was contained in the investigational vaccine as a carrier protein. Anti-tetanus antibodies were measured by electrochemiluminescent (ECL) assay. The captured antibodies were then detected using a sulfotag-conjugated anti-human immunoglobulin (Ig)G conjugate.
Time Frame: Pre-dose Day 0 and Day 30 post-dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: International units/milliliter (IU/mL)
Arm/Group | MenACYW Conjugate Vaccine
Number analyzed (Participants) | 287
International units/milliliter (IU/mL)
  Day 0 (pre-dose): number analyzed (Participants) | 286
  Day 0 (pre-dose) | 0.040 [0.033 to 0.049]
  Day 30 (post-dose) | 0.429 [0.291 to 0.631]

5. Primary Outcome: Percentage of Participants Who Achieved Seroprotective Levels
Description: Seroprotective levels defined as antibody titers >= 0.01 IU/mL and >= 0.1 IU/mL of antibody concentrations to tetanus toxoid. Tetanus toxoid was contained in the investigational vaccine as a carrier protein. Anti-tetanus antibodies were measured by ECL assay. The captured antibodies were then detected using a sulfotag-conjugated anti-human IgG conjugate. Percentages are rounded off to the tenth decimal place.
Time Frame: Pre-dose Day 0 and Day 30 post-dose
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW Conjugate Vaccine
Number analyzed (Participants) | 287
percentage of participants
  Day 0 (pre-dose): >=0.01 IU/mL: number analyzed (Participants) | 286
  Day 0 (pre-dose): >=0.01 IU/mL | 87.8 [83.4 to 91.3]
  Day 0 (pre-dose): >=0.1 IU/mL: number analyzed (Participants) | 286
  Day 0 (pre-dose): >=0.1 IU/mL | 28.3 [23.2 to 33.9]
  Day 30 (post-dose): >=0.01 IU/mL | 93.0 [89.4 to 95.7]
  Day 30 (post-dose): >=0.1 IU/mL | 56.8 [50.8 to 62.6]

6. Primary Outcome: Number of Participants With Unsolicited Systemic Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE is an observed AE that does not fulfill the conditions of solicited reactions [i.e.pre-listed in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination].
Time Frame: Within 30 minutes post-dose
Population: The Safety analysis set (SafAS) consisted of participants who had received at least 1 dose of the study vaccine and had any safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW Conjugate Vaccine
Number analyzed (Participants) | 288
Participants | 0

7. Primary Outcome: Number of Participants With Solicited Injection Site Reactions and Systemic Reactions
Description: All noxious and unintended responses to a study vaccine related to any dose was considered adverse reactions (AR). A solicited reaction is an "expected" AR (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRB. An injection site reaction is an AR at and around the injection site. Injection site reactions are commonly inflammatory reactions. They were considered to be related to the study vaccine administered. Systemic reactions were all ARs that were not injection or administration site reactions and included systemic manifestations such as headache, fever, as well as localized or topical manifestations that are not associated with the vaccination or administration site.
Time Frame: Up to 7 days post-dose
Population: The SafAS consisted of participants who had received at least 1 dose of the study vaccine and had any safety data available. Only those participants with data collected are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW Conjugate Vaccine
Number analyzed (Participants) | 287
Participants
  Solicited injection site reaction | 39
  Solicited systemic reaction | 59

8. Primary Outcome: Number of Participants With Unsolicited Non-Serious Adverse Events
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE is an observed AE that does not fulfill the conditions of solicited reactions (i.e. pre-listed in the CRB in terms of diagnosis and/or onset window post-vaccination).
Time Frame: Up to Day 30 post-dose
Population: The SafAS consisted of participants who had received at least 1 dose of the study vaccine and had any safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW Conjugate Vaccine
Number analyzed (Participants) | 288
Participants | 41

9. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAEs is defined as any untoward medical occurrence, at any dose that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, or other important medical event.
Time Frame: From Day 0 up to end of study, approximately 44 days
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW Conjugate Vaccine
Number analyzed (Participants) | 288
Participants | 6

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from Day 0 up to end of study, approximately 44 days. All-cause mortality (death) was collected from signing of the informed consent form to the end of safety follow-up, a maximum of 35 months.
Description: Analysis was performed on SafAS population.
Groups:
- MenACYW: Participants received a single dose of meningococcal polysaccharide [Serogroups A, C, W and Y (MenACYW conjugate vaccine)] 0.5 mL IM injection on Day 0.
Arm/Group | MenACYW
All-Cause Mortality (participants affected / at risk) | 1/288
Serious Adverse Events (participants affected / at risk) | 6/288
Other Adverse Events (participants affected / at risk) | 69/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACYW (N=288)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypertensive Encephalopathy (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACYW (N=288)
Injection Site Pain (General disorders) | 40 (41)
Malaise (General disorders) | 27 (27)
Myalgia (Musculoskeletal and connective tissue disorders) | 38 (38)
Headache (Nervous system disorders) | 48 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT03869866/Prot_002.pdf
  • Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT03869866/SAP_003.pdf